CLINICAL TRIAL: NCT01847339
Title: A Study of Epidural Bupivacain-soaked Absorbable Gelatin Sponge on Post-operative Pain in Lumbar Laminectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 13-183
Record Dates: First submitted 2013-05-02; First posted 2013-05-06 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lumbar Laminectomy
MeSH Terms: interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine soaked sponges (Experimental): Patients will be randomized using a reproducible set of computer-generated random numbers. In study group a 1 square centimeter piece of absorbable gelatin sponge will be soaked in the bupivacaine solution %0.25 and then will be placed by the surgeon in the epidural space before final closure
  Interventions: Drug: bupivacaine
- saline soaked sponges (Placebo Comparator): Patients will be randomized using a reproducible set of computer-generated random numbers. In study group a 1 square centimeter piece of absorbable gelatin sponge will be soaked in saline solution and then will be placed by the surgeon in the epidural space before final closure.
  Interventions: Other: saline solution

INTERVENTIONS:
Drug: bupivacaine — In study group a 1 square centimeter piece of absorbable gelatin sponge will be soaked in the bupivacaine solution %0.25 and then will be placed by the surgeon in the epidural space before final closure.
  Arms: bupivacaine soaked sponges
Other: saline solution — In study group a 1 square centimeter piece of absorbable gelatin sponge will be soaked in the saline solution and then will be placed by the surgeon in the epidural space before final closure
  Arms: saline soaked sponges

SUMMARY:
The effective relief of pain is of paramount importance to anyone treating patients undergoing surgery. Post-operative pain increases the possibility of post-surgical complications, raises the cost of medical care, and most importantly, interferes with recovery and return to normal activities of daily living. Therefore pain control is essential in the management of patients undergoing spinal surgery.Parenteral administration of narcotics has been the mainstay for postoperative pain relief in patients undergoing laminectomy and discectomy. Epidural and intrathecal opioids are also effective means of pain control in several major surgical interventions including spinal surgery. However, some of the side effects have limited their widespread use (eg, late-onset respiratory depression). Therefore, alternative measures of pain control including infiltration of paraspinal musculature with local anesthetics have been investigated with conflicting results. In situations such as laminectomies, where the epidural space is exposed as part of the surgical procedure, the application of absorbable gelatin sponge soaked in local anesthetics appears to be an alternative for providing postoperative analgesia. By investigating the probable analgesic effects of this method the investigators may relieve post laminectomy pain with minimal side effects and also costs.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I or III
* scheduled to undergo lumbar laminectomy

Exclusion Criteria:

* Patients who are younger than 18 years of age
* pregnant
* spinal or lateral stenosis
* previous intervertebral disc surgery at that level
* patients with history of chronicity (symptoms >6 months duration) or coexisting medical conditions such as substance abuse or withdrawal, hyperthyroidism, anxiety disorder, affective disorder, hepatic or renal impairments

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02-12 (Actual)

PRIMARY OUTCOMES:
reported post operative pain | Day 1
  We will test the hypothesis, that the bupivacaine-soaked sponge reduces postoperative pain or reduces opioid consumption in patients undergoing spinal surgery.
recorded opioid consumption | Day 1
  We will test the hypothesis, that the bupivacaine-soaked sponge reduces postoperative pain or reduces opioid consumption in patients undergoing spinal surgery.

SECONDARY OUTCOMES:
reported pain | Day 1
  Bupivacaine epidural sponge increases the time from the end of the operation until the patient requested supplementation of analgesic.
reported side effects | Day 1
  We will also evaluate side effects of this method of analgesia such as sedation, urinary retention, hypotension, respiratory depression, nausea, vomiting and extremity weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Firoozbakhsh, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States